CLINICAL TRIAL: NCT00788385
Title: Multi-Center Study of ShuntCheck
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: NeuroDx Development (Industry)
Responsible Party: Fred Fritz, Neuro Diagnostic Devices
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: NDX01-22-2001
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Blocked Ventricular Shunts
Keywords: Hydrocephalus; High Pressure; Shunt Blockage
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ShuntCheck test

SUMMARY:
Multi-Center Study of ShuntCheck

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

Ages: 1 Month to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)